CLINICAL TRIAL: NCT01398306
Title: Biomarkers for Angiogenesis in Renal Cell Carcinoma and Neuro-endocrine Tumours.
Acronym: BANN
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: 230520112
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Carcinoma; Carcinoma, Renal Cell; Neuroendocrine Tumors; Carcinoid Tumor; Pancreatic Islet Cell Tumors
Keywords: Angiogenesis Inhibitors; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Adenocarcinoma; Kidney Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Kidney Diseases; Angiogenesis Inducing Agents; Biological Markers
MeSH Terms: conditions — Carcinoma; Carcinoma, Renal Cell; Neuroendocrine Tumors; Carcinoid Tumor; Adenoma, Islet Cell; Neoplasms, Glandular and Epithelial; Neoplasms by Histologic Type; Neoplasms; Adenocarcinoma; Kidney Neoplasms; Urologic Neoplasms; Urogenital Neoplasms; Neoplasms by Site; Kidney Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — 2 x 10mL whole blood, stored as platelet rich and platelet poor plasma.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group A: Patients with clear cell renal cell carcinoma with metastases.
  Interventions: Other: Blood sampling by vena punction.
- Group B: Patients with low grade neuro-endocrine tumours with metastases.
  Interventions: Other: Blood sampling by vena punction.

INTERVENTIONS:
Other: Blood sampling by vena punction. — We obtain 10mL blood of the patients. The blood is obtained twice: once with angiogenesis inhibitors or mTOR inhibitors, and once without.

SUMMARY:
The primary objective of this study is to analyse the concentration dopamine and serotonin in thrombocytes of patients with renal cell carcinoma and neuro-endocrine tumours compared to the concentrations of these catecholamines in healthy volunteers. The concentration dopamine and serotonin in thrombocytes with and without medication will also be evaluated.

DETAILED DESCRIPTION:
* To analyse the concentration catecholamines in thrombocytes of patients with clear cell renal cell carcinoma and low grade neuroendocrine tumours.
* To compare these concentrations with the concentrations catecholamines in thrombocytes of healthy controls.
* To analyse the concentration catecholamines in thrombocytes of patients with clear cell renal cell carcinoma and patients with low grade neuroendocrine tumours with and without medication.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years old or older.
* Patients with clear cell renal cell carcinoma with metastases or patients with a low-grade neuro-endocrine tumor with metastases.
* Written informed consent

Exclusion Criteria:

* Use of L-dopa or SSRI.
* Patients with a second primary malignancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with clear cell renal cell carcinoma with metastases and patients with low grade neuroendocrine tumours with metastases.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-07; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Difference in concentrations DA and 5-HT in thrombocytes of patients with clear cell renal cell carcinoma and healthy controls, and patients with low grade neuroendocrine tumours and healthy controls. | one year

SECONDARY OUTCOMES:
Difference in concentrations DA and 5-HT in thrombocytes of patients with clear cell renal cell carcinoma and low grade neuroendocrine tumours with and without medication. | one year

CONTACTS AND LOCATIONS:
Overall Officials: Sjoukje F. Oosting, MD, Study Chair — University Medical Center Groningen; Marloes A.M. Peters, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands